Humira® for subcutaneous use only

Special drug-use survey

-Long-term survey on Crohn's disease-

Final report
Statistical Analysis Plan

-Ver. 1.0-

Prepared on Apr 02, 2018

1. Approval

Entruster

Company name AbbVie GK

Approved by Post-marketing Surveillance Supervisor Seal

Date of approval MMM, DD, YYYY

Approved by Medical Supervisor Seal

Date of approval MMM, DD, YYYY

Approved by Safety Management Supervisor Seal

Date of approval MMM, DD, YYYY

Approved by Survey Planning Physician Seal

Date of approval MMM, DD, YYYY

Approved by Statistical Analysis Supervisor Seal

Date of approval MMM, DD, YYYY

Entruster

Company name Eisai Co., Ltd.

Approved by Drug Development Planning: Statistical Analysis Supervisor Seal

Date of approval MMM, DD, YYYY

Entrustee

Company name A2 Healthcare Corporation

Approved by Statistical Analysis Project Leader Seal

Date of approval MMM, DD, YYYY

# Table of Contents

| 1. Prep | paration/revision history | 9 |
|---------|--------------------------------------------------------|----|
| 2. Def | initions of terms and abbreviations | 9 |
| 3. Obj | ective of this statistical analysis plan | 10 |
| 3.1. | Objective of developing this statistical analysis plan | 10 |
| 4. The | survey outline | 10 |
| 4.1. | Survey objective | 10 |
| 4.2. | Survey plan | 10 |
| 4.3. | Target sample size for the survey | 10 |
| 5. Item | ns to be analyzed and the methods | 11 |
| 5.1. | Items for analysis | 11 |
| 5.2. | Analysis method | 11 |
| 6. Pres | sence/absence of analysis and its schedule | 11 |
| 7. Soft | twares/dictionary used for analysis | 12 |
| 7.1. | Statistical analysis and listing softwares | 12 |
| 7.2. | Dictionary for use | 12 |
| 8. The | definition of the groups used for analysis | 13 |
| 9. Gen | eral agreement items for analysis | 14 |
| 9.1. | Handling of missing data | 14 |
| 9.2. | Descriptive statistics | 15 |
| 9.3. | Display digit for figures | 15 |
| 9.4. | Figure display rule | 16 |
| 9.5. | Statistical test method | 16 |
| 9.6. | Significant level | 16 |
| 10. Der | ivation and calculation methods for data | 17 |
| 10.1. | General | 17 |
| Nun | nber of sites for this survey | 17 |
| The | first administration date of Humira. | 17 |
| The | final administration date of Humira | 17 |
| Day | rs to the final administration date of Humira | 18 |
| Tota | al exposure period (in years) | 18 |
| Disc | continued patients | 18 |
| Rea | son for discontinuation | 18 |
| Dea | th cases | 18 |
| Ped | iatrics | 18 |
| The | elderly | 18 |
| Pres | sence/absence of complications | 19 |
| Con | nplication/Hepatic function disorder | 19 |

| Complication/Renal impairment | 19 |
|--------------------------------------------------------------------|----|
| Complication/Blood disorder | 19 |
| Complication/Respiratory disorder | 19 |
| Complication/others | 19 |
| Intestinal complications | 20 |
| Non-intestinal complications | 20 |
| Presence/absence of medical history | 20 |
| Medical history: tuberculosis | 20 |
| Medical history: non-tuberculous mycobacteriosis | 20 |
| Medical history: interstitial pneumonia | 20 |
| Medical history: bronchitis bacterial | 20 |
| Medical history: aplastic anaemia | 21 |
| Medical history: pancytopenia | 21 |
| Medical history: malignant tumour | 21 |
| Patients with an hepatitis B virus infection | 21 |
| Presence/absence of administration of anti-hepatitis B virus agent | 21 |
| Presence/absence of allergy history | 21 |
| Presence/absence of smoking history | 22 |
| Details of smoking history | 22 |
| Administration status | 22 |
| Administration status (total number of dosing, total dose) | 23 |
| Patients with self-administration | 23 |
| Age | 23 |
| Indication | 23 |
| Tuberculin test | 24 |
| QuantiFeron test | 24 |
| Chest X ray test | 24 |
| Thoracic CT test | 24 |
| Imaging procedure | 24 |
| Tuberculosis test | 24 |
| Patients subject to AAA measurement | 24 |
| Patients of contraindications | 24 |
| Patients who developed an infection | 24 |
| Patients who developed malignant tumour | 24 |
| Duration of illness (in years) | 24 |
| Concomitant medication | 25 |
| Concomitant medication: aminosalicylic acid products | 26 |
| Concomitant medication: corticosteroid | 26 |

| | Concomitant medication: immunosuppressant | 26 |
|---|---|---|
| | Concomitant medication: antibiotics | 26 |
| | Concomitant medication: others | 26 |
| | Prior medication: TNFα drug | 26 |
| | Prior medications | 26 |
| | Prior medication: aminosalicylic acid products | 27 |
| | Prior medication: corticosteroid | 27 |
| | Prior medication: immunosuppressant | 27 |
| | Prior medication: antibiotics | 27 |
| | Prior treatment | 27 |
| | Prior treatment: surgery | 27 |
| | Prior treatment: granulocyte and monocyte adsorption apheresis (GCAP) | 27 |
| | Prior treatment: enteral nutrition therapy | 27 |
| | Prior treatment: intravenous nutrition therapy | 27 |
| | Concomitant therapy | 27 |
| | Concomitant therapy: surgery | 28 |
| | Concomitant therapy: GCAP | 28 |
| | Concomitant therapy: enteral nutrition therapy | 28 |
| | Concomitant therapy: intravenous nutrition therapy | 28 |
| | Work condition | 28 |
| 1 | 0.2. Safety analysis | 28 |
| | Adverse event | 28 |
| | Seriousness of adverse events | 28 |
| | Causal relationship of adverse events | 29 |
| | Outcome of adverse events | 29 |
| | Days from the first administration date of Humira to the adverse-event onset date | 29 |
| | Days from the adverse-event onset date to the outcome confirmation date (recovered | d or |
| | recovering) | 29 |
| | Incidence of adverse reactions, incidence of serious adverse reactions, incidence of adverse | erse |
| | events, incidence of serious adverse events | 30 |
| 1 | 0.3. Effectiveness analysis | 30 |
| | Remission. | 30 |
| | WPAI | 30 |
| 11. | How to stratify data | 32 |
| 12. | Data handling at test/assessment periods | 35 |
| 1 | 2.1. Assessment period for CDAI, WPAI, CRP and non-intestinal conditions | 35 |
| 1 | 2.2. Assessment period of endoscopy results | 35 |
| 1 | 2.3. Assessment period for the administration status of Humira | 36 |

| 1 | 2.4. | Assessment period for the onset status of adverse reactions | 36 |
|---|---|---|---|
| 1 | 2.5. | Assessment period for the continued administration of Humira | 37 |
| 13. | Charts | to be generated (chart No., chart name) | 37 |
| 1 | 3.1. | General | 37 |
| | "1.1.1 | Case structure chart" | 37 |
| | "1.1.2 | Case structure chart on patients in the effectiveness analysis group" | 37 |
| | "1.2 N | lumber of sites surveyed and number of patients surveyed (patients in the safety anal | lysis |
| | group) | " | 38 |
| | "1.1.3 | Progress in survey forms" | 38 |
| | "1.3 A | a list of the patients excluded from the safety analysis and the patients excluded from | the |
| | effecti | veness analysis (including the reason for exclusion)" | 38 |
| | "1.3.1 | Excluded patients (aggregation by reason)" | 39 |
| | "1.4 A | list of patients (adverse event + search flag)" | 39 |
| | "1.4.1 | A list of adverse events" | 40 |
| | "1.4.2 | A list of death cases" | 40 |
| | "1.4.3 | A list of patients aged 18 years or younger" | 41 |
| | "1.5 A | dministration status of Humira (dosage and administration)" | 41 |
| | | Administration status of Humira (dosing frequency, dose) | |
| | | Administration status of Humira (period)" | |
| | | Continuation rate of Humira" | |
| | "1.7 A | dministration status of Humira (discontinuation of administration)" | 42 |
| | "1.7.1 | Administration status of Humira (reason for discontinuation other reasons) | 43 |
| | "1.7.2 | Administration status of Humira (a list of reasons for discontinuation other reasons)". | 43 |
| | | Distribution status of patient backgrounds" | |
| | | Distribution status of self-administration" | |
| | "1.16 | A list of patients with AAA measured | |
| 1 | 3.2. | Safety | |
| | | list of the onset status of serious adverse events (Attachment Form 10)" | |
| | | list of target-patient summary (Attachment Form 3)" | |
| | | .1 A list of the onset status of adverse reactions (priority survey items)" | |
| | | 2 A list of the onset status of adverse events (priority survey items)" | |
| | | A list of the onset status of the priority survey items per 100 patient-year" | |
| | | A list of the onset status of adverse reactions with/without self-administration" | |
| | | A list of the onset status of adverse reactions with/without self-administration" | |
| | | ncidence of adverse reactions per onset period (serious)" | |
| | | ncidence of adverse reactions per set period" | |
| | | Incidence of adverse reactions (serious adverse reactions/adverse reactions) | - |
| | backgr | round factor" | 50 |

| "2.9.xx Incidence of adverse reactions per background factor and seriousness"51 |
|---|
| "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per |
| seriousness" |
| "2.14.1 Incidence of adverse reactions with/without renal impairment and per seriousness"52 |
| "2.15.1 Incidence of adverse reactions per seriousness in pediatrics and non-pediatrics"52 |
| "2.16.1 Incidence of adverse reactions per seriousness in the elderly and non-elderly patients" |
| 53 |
| "2.17.1 A list of the onset status of adverse reactions/infections in this survey"53 |
| "2.17.2 A list of the onset status of adverse reactions/infections not in the follow-up period"53 |
| "2.17.3 A list of the onset status of adverse reactions/infections in this survey (patients excluded |
| from the safety analysis)" |
| "2.19 A list of the onset status of adverse events in this survey"54 |
| "2.20 A list of the onset status of adverse reactions (all cases)"54 |
| 3.3. Effectiveness |
| "3.1 CDAI remission rate at the final assessment (CDAI<150)"55 |
| "3.2.1.1 Changes in Crohn's disease activity index (CDAI) since the administration was started |
| (Observed Case)" |
| "3.2.1.2 Changes in Crohn's disease activity index (CDAI) since the administration was started |
| (Observed Case)" |
| "3.2.2.1 Changes in the remission rate at each point (CDAI<150) (Observed Case)"56 |
| "3.2.2.3 Changes in the remission rate at each point (CDAI<150) (Observed Case)"56 |
| "3.2.4.2 Endoscopy results during administration (small intestine: active phase/remission phase)" |
| 57 |
| "3.2.5.2 Endoscopy results during administration (large intestine: active phase/remission phase)" |
| 57 |
| "3.2.5.3 Endoscopy results during administration (remission phase in both small and large |
| intestines)" |
| "3.2.6.2 Changes in WPAI:CD since the administration was started (Observed Case)"58 |
| "3.2.7.2 Changes in CRP level since the administration was started (Observed Case)"58 |
| "3.2.7.3 Remission rate at the final assessment in patients who achieved a remission of CDAI at |
| Week 4 of administration" |
| "3.2.8 Subsequent changes in the conditions of patients with non-intestinal conditions observed |
| at the first administration (Observed Case)" |
| "3.4.1 Aggregation for effectiveness per patient background factor (CDAI)" |

## 1. Preparation/revision history

| Version<br>No. | Date of preparation/revision | Prepared/revised by | Reasons |
|---|---|---|---|
| 1.0 | APR 02,2018 | | First version |

## 2. Definitions of terms and abbreviations

The terms and abbreviations used in this analysis plan are as follows:

| Term and abbreviation | Definition |
|---|---|
| Adverse event | Any untoward or unintended symptoms (including abnormal laboratory findings), condition or illness which are not always related to Humira. |
| Adverse events in the safety analysis period | Adverse events which occur from the first administration date of Humira through Week 160 of administration (Day 1 + 1120). Note that if a date is not provided, it should also be included in the period for analysis. |
| Adverse events not in<br>the safety analysis<br>period | Adverse events which occur prior to the first administration date of Humira or beyond Week 160 of administration (Day 1 + 1120). |
| Adverse reaction | Adverse events for which the causal relation with Humira cannot be ruled out. |
| Adverse reactions in the safety analysis period | Adverse events which occurred in the safety analysis period and for which the causal relation with Humira cannot be ruled out. |
| Adverse reactions not in the safety analysis period | Adverse events which occurred not in the safety analysis period and for which the causal relation with Humira cannot be ruled out. |
| MedDRA/J | Medical Dictionary for Regulatory Activities / Japanese edition |
| SOC | System Organ Class in MedDRA/J |
| PT | Preferred Terms in MedDRA/J |
| LLT | Lowest Level Terms in MedDRA/J |
| CDAI Crohn's Disease Activity Index | |
| WPAI | Work Productivity and Activity Impairment Questionnaire : Crohn's Disease |
| CRP | C-reactive protein |
| GB | Green book. Guide on re-examination |

#### 3. Objective of this statistical analysis plan

#### 3.1. Objective of developing this statistical analysis plan

This statistical analysis plan aims at planning in advance the items regarding the statistical analysis activities which are conducted in accordance with the protocol of "Special drug-use survey for Humira® for subcutaneous use only (the long-term survey on Crohn's disease)" (hereinafter referred to as "this survey"). This is a survey conducted in accordance with GPSP Ministerial Ordinance, and is a document used to prepare the regulatory report of Humira's special drug-use survey and application documents for re-examination.

#### 4. The survey outline

#### 4.1. Survey objective

The survey aims to collect information on the safety (especially, the onset status of malignant tumour and serious infections) and the effectiveness in Crohn's-disease patients who used Humira<sup>®</sup> for subcutaneous use only (hereinafter, this drug) and to review and discuss the safety and effectiveness.

<Priority survey items>

Onset status of malignant tumour, serious infection, etc.

#### 4.2. Survey plan

The target patients for this survey should satisfy the following items when the survey is started:

- [1] A Crohn's-disease patient who is a suitable candidate for the indication, dosage and administration of Humira
- [2] A patient with no malignant tumour in medical history and as complication.
- [3] A patient who is not treated with this drug today

#### 4.3. Target sample size for the survey

500 patients

The incidence of malignant tumour when this drug was approved was 1.1% (1/90) in the domestic clinical study and 1.1% (16/1459) in the overseas clinical study in Crohn's disease-patients, showing that malignant tumour occurred in approximately 1.0% of the patients both in Japan and overseas. Therefore, we have a sample size of approximately 300 patients for this survey to detect at least one patient who develops malignant tumour with a power of 95%. We are going to register 500 patients in view of possible withdrawals and dropouts in the follow-up period.

## 5. Items to be analyzed and the methods

#### 5.1. Items for analysis

- 1) Items regarding patient composition
  - [1] The number of registered patients
  - [2] The number of patients whose survey form was collected
  - [3] The number of patients in the safety analysis group
  - [4] The number of patients in the effectiveness analysis group
- 2) Items regarding safety
  - [1] A list of the onset status of adverse reactions/malignant tumour/infections
  - [2] Possible factors which may affect the safety
    - · Incidence of adverse reactions per patient background, etc.
  - [3] The onset status of adverse events
    - · A list of the onset status of serious adverse events
  - [4] The administration-error status at self-administration
- 3) Items regarding effectiveness

CDAI, WPAI:CD, Endoscopy, CRP

4) Others

We are going to stratify and analyze malignant tumour, tuberculosis, serious infections, etc.

#### 5.2. Analysis method

Appropriate tests including  $\chi^2$  test are employed for analysis, depending on the analysis-data scale and the characteristics.

#### 6. Presence/absence of analysis and its schedule

| Analysis objective | The survey's reporting interval and the deadline of re-examination |
|---|---|
| Final report | From November, 2011 to March, 2017 |

## 7. Softwares/dictionary used for analysis

## 7.1. Statistical analysis and listing softwares

The softwares and their versions for use are as follows:

| | Software and version |
|---|---|
| OS | We use Microsoft Windows 7 or a more recent version. |
| Statistical analysis software | We use SAS Ver. 9.2 or a more recent version. |
| Listing software | We use Microsoft Excel 2010 or a more recent version. |

## 7.2. Dictionary for use

The dictionaries used for the names of adverse events, complications, and drugs are as follows:

| Item | Dictionary and its version | Remarks |
|---|---|---|
| Types of adverse events<br>and adverse<br>reactions/infections | Medical Dictionary for Regulatory Activities / Japanese edition (MedDRA/J 20.1) | <ul> <li>They are classified into a System Organ Class (SOC) and the appropriate term among the preferred terms (PT) is selected for description.</li> <li>SOC is displayed in accordance with the international agreement.</li> <li>The MedDRA/J version used will be provided in a blank space.</li> </ul> |
| Drug name (concomitant medication) | Iyakuhinmei Data File (IDF) *An appropriate version is applied, depending on the analysis period. | <ul> <li>A 7-digit code is used, in principle, when concomitant medications are counted per product.</li> <li>Give a priority to the lowest level codes when using codes for the list of concomitant medications (including Re-examination Attachment Form 3).</li> </ul> |

## 8. The definition of the groups used for analysis

| Name of group | Definition |
|---|---|
| Patients for registration | Patients whose registration was fixed. |
| Patients whose survey form was locked | The patients for whom the survey form was locked. |
| Patients whose survey<br>form was yet to be<br>locked | Patients whose survey form was yet to be locked |
| Patients excluded from the safety analysis group The patients whose survey form has been locked and who criteria of the patients excluded from the safety analysis "Document for Inclusion/exclusion of patients (for final the criteria to exclude patients from the safety analysis group) | |
| Patients in the safety analysis group | The remaining patients after the patients excluded from the safety analysis group are removed from the patients whose survey form was locked. |
| Patients excluded from<br>the effectiveness analysis<br>group | Patients who satisfy the exclusion criteria of the effectiveness analysis. See "Document for Inclusion/exclusion of patients (for final reporting)" for the criteria to exclude patients from the effectiveness analysis group. |
| Patients in the effectiveness analysis group | The remaining patients after those excluded from the effectiveness analysis group are removed from the patients in the safety analysis group. |

## 9. General agreement items for analysis

## 9.1. Handling of missing data

The relevant item's definition at Chapter 10 or thereafter defines how to impute data. In addition, for date imputation, follow the table below to impute the dates.

| Tession | Entry data | | Dates after | | |
|---|---|---|---|---|---|
| Item | year | month | day | imputation | Replacement |
| Chest X ray,<br>Thoracic CT, other | 2018 | 1, | null | January 1,<br>2018 | If a date is null, regard it as the first day of the month. |
| imaging, Tuberculin<br>test, QuantiFeron | 2018 | 1 | -97 | January 1,<br>2018 | If a date is unknown, regard it as the first day of the month. |
| test, endoscopy | 2018 | 1 | The first<br>10 days<br>of a<br>month | January 1,<br>2018 | If a date is any of the first 10 days of a month, regard it as the first day of the month. |
| CRP | 2018 | 1 | null | null | If the date is null, it is regarded as null. |
| | 2018 | 1 | The end of a month | January<br>31, 2018 | If the date is "the end of month", replace it with the actual end date of the applicable month. |
| CDAI | null | 1 | 1 | null | If a year is null, it is regarded as null. |
| General (including the items above and | -97 | -97 | <del>-</del> 97 | null | If a year, a month and a date are all unknown, they are regarded as null. |
| WPAI) | null | null | null | null | If a year, a month and a date are all null, they are regarded as null. |
| | 2018 | -97 | -97 | null | If a month and a date are unknown, they are regarded as null. |
| | 2018 | null | null | null | If a month and a date are null, they are regarded as null. |

## 9.2. Descriptive statistics

The following will be calculated for categorial data and quantitative data.

| Data type | Item to be calculated |
|---|---|
| Categorical data | Number of patients, percentage, etc. When the percentage is calculated, the number of patients of "unknown/not provided" is included in the denominator. Chapter 13 stipulates the details regarding the setting of denominators. The patients of "unknown" and "not provided" are excluded in the statistical test. |
| Quantitative data | Summary statistics: number of cases, mean, standard deviation, median, minimal value, maximal value, 1st quartile value, and 3rd quartile value |

## 9.3. Display digit for figures

The display digit for figures is as follows:

| Type of figure | Display digit |
|---|---|
| Mean, standard<br>deviation, median, 1st<br>quartile value, 3rd<br>quartile value, 95%<br>confidence interval | The figure in the significant digit + 2 digits of data is rounded off to the figure in the significant digit of data + 1 digit for display. |
| Minimal value,<br>maximal value | The same number of digits is used for the significant digit of data. |
| Number of patients | Displayed as a whole number |
| Percentage | The figure is rounded off to the nearest one decimal place for display. When figures for Attachment Form 2, incidences of adverse events, etc are rounded off to two decimal places, the details are specified in the chart layout. |
| p value | Round the 5 decimal places down to the 4 decimal places. When the figure is smaller than 0.0001, display it as <0.0001 across the board. |
| Significant digit | The figure for duration of illness should be displayed with the significant digit rounded to the one decimal place. For others, the display digit of data should be the significant digit. As for CRP, the summary statistics except the number of patients should be rounded off to two decimal places. |

## 9.4. Figure display rule

| Case | Display rules |
|----------------|---------------|
| If a figure is | Hyphen "-" |
| incalculable | |

#### 9.5. Statistical test method

The test does not include the classification of unknown/not provided. In principle, the first layer is subjected to the intersegmental test of classified data. Multiplicity is not adjusted.

## 9.6. Significant level

In principle, the significant level is 5%, two-tailed. p<0.05 (<5%) shall be considered significant.

## 10. Derivation and calculation methods for data

# 10.1. General

| Data name | Derivation and calculation methods |
|---|---|
| Number of sites for this survey | Aggregate the number with DCF code. |
| The first administration | It shall be the oldest date among the dates described in "the |
| date of Humira | administration status of Humira" in the survey form. |
| The final administration date of Humira | Do not use for analysis the record of the first administration date of Humira + 1092 days < the first administration date among the data described in "the administration status of Humira" in the survey form. The final administration date of Humira shall be the most recent date among the final administration dates imputed in the following [1] to [4]: [1] Sort data in the order of "the first administration date" of "the administration status of Humira", dosing frequency and description. [2] If the final date is provided, there is no check on the checkbox of "continued", and the final administration date can be identified, select the date described as the final administration date. If the final date is not described, the checkbox of "continued" is checked, and the final administration date cannot be identified, follow the below: The final record: Impute the first administration date of Humira + 1092 days on the final administration date. Other than the final record: Impute the first administration date. Seven though the final dates are described, but the final administration date is incomplete and cannot be identified, follow the below: If the year and month are described but the date is unknown, impute the final date of the month as the final administration date. If the year is described and the month and date are unknown, impute the final date of the year as the final administration date. If the next record has already been generated and the first administration date of the next record comes earlier than the imputed date, impute the first administration date of the next record comes earlier than the imputed date, impute the first administration date of the next record comes earlier than the imputed date, impute the first administration date of the next record comes earlier than the imputed date, impute the first administration date of the next |

| Data name | Derivation and calculation methods |
|---|---|
| | record - 1 day for the final administration date. |
| | Of note, if the final administration date is provided in the record where<br>the final administration date of Humira has been identified according to |
| | the above rule and the "continued" checkbox is checked, follow the below: |
| | <ul> <li>If the described final administration date &gt; the final administration date imputed according to the above rule, select the imputed final administration date as the final administration date of Humira for the patient.</li> <li>If the described final administration date &lt;= the final</li> </ul> |
| | administration date imputed according to the above rule, select<br>the described final administration date as the final<br>administration date of Humira for the patient. |
| | If the first administration date of Humira + 1092 days < the final administration date of Humira imputed according to the above rule, select the first administration date of Humira + 1092 days as the final |
| | administration date of Humira. |
| Days to the final<br>administration date of<br>Humira | The final administration date of Humira - the first administration date of Humira + 1 |
| Total exposure period (in years) | (Days to the final administration date of Humira + 28) / 364 |
| Discontinued patients | <ul> <li>Patients whose final administration date of Humira comes before the first administration date of Humira + 1064 (Week 152)</li> <li>Patients with a washout period with 60 days or longer.</li> <li>*The final administration date of Humira should be the administration date right before the washout of ≥60 days starts.</li> </ul> |
| Reason for discontinuation | When a reason for discontinuation is described in the survey form, it is defined as 'with' reason for discontinuation. When no such description is found, it is defined as an "unknown/not provided". |
| Death cases | At least a piece of data on "death" is found as the outcome of the adverse events during the safety analysis period. |
| Pediatrics | Patients aged <15 years |
| The elderly | Patients aged ≥65 years |

| Data name | Derivation and calculation methods |
|---|---|
| Presence/absence of | When complication data are contained in the survey form, it should be |
| | classified as "with complications". When the description in the survey |
| | form is not clear enough (when the check of with/without complications |
| complications | is not assessable or when multiple checkboxes are checked), it should be |
| | 'unknown" while no description should be 'not provided'. Other cases |
| | are "no complications". |
| | When liver-disorder data are contained in "171210 Complications.xlsx", |
| | it should be classified as "with hepatic function disorder". When the |
| Complication/Hepatic | description in the survey form is not clear enough (when the check of |
| function disorder | with/without complications is not assessable or when multiple |
| | checkboxes are checked), it should be 'unknown' while no description |
| | should be 'not provided'. Other cases are "no hepatic function disorder". |
| | When renal-disorder data are contained in "171210 |
| | Complications.xlsx", it should be classified as "with renal impairment". |
| Complication/Renal | When the description in the survey form is not clear enough (when the |
| impairment | check of with/without complications is not assessable or when multiple |
| | checkboxes are checked), it should be 'unknown' while no description |
| | should be 'not provided'. Other cases are "no renal impairment". |
| | When blood-disorder data are contained in "171210 |
| | Complications.xlsx", it should be classified as "with blood disorder". |
| Complication/Blood | When the description in the survey form is not clear enough (when the |
| disorder | check of with/without complications is not assessable or when multiple |
| | checkboxes are checked), it should be 'unknown" while no description |
| | should be 'not provided'. Other cases are "no blood disorder". |
| | When respiratory-disorder data are contained in "171210 |
| | Complications.xlsx", it should be classified as "with respiratory |
| C 1: .: /P : . | disorder". When the description in the survey form is not clear enough |
| Complication/Respirato | (when the check of with/without complications is not assessable or when |
| ry disorder | multiple checkboxes are checked), it should be 'unknown" while no |
| | description should be 'not provided'. Other cases are "no respiratory |
| | disorder". |
| | When other data are contained in "171210 Complications.xlsx", it |
| | should be classified as "with others". When the description in the survey |
| Complication/others | form is not clear enough (when the check of with/without complications |
| | is not assessable or when multiple checkboxes are checked), it should be |
| | 'unknown" while no description should be 'not provided'. Other cases |

| Data name | Derivation and calculation methods |
|---|---|
| | are "no others". |
| E 8 88 E | Classify the complications as mentioned in the presence/absence of |
| | intestinal-complications column of survey form. |
| Intestinal | Of note, if the presence/absence check is not assessable or multiple |
| complications | checkboxes are checked, it should be classified into 'unknown', while |
| | no description should be 'not provided'. |
| | Classify the complications as mentioned in the presence/absence of non |
| A9 (610) 06 N | intestinal-complications column of survey form. |
| Non-intestinal | Of note, if the presence/absence check is not assessable or multiple |
| complications | checkboxes are checked, it should be classified into 'unknown', while |
| | no description should be 'not provided'. |
| | When medical-history data are contained in the survey form, it should |
| Presence/absence of | be classified as "with medical history". When the checkbox of 'medical |
| medical history | history unknown' is checked, it should be 'unknown' while no |
| | description should be 'not provided'. Others are "no medical history". |
| | When medical-history data on tuberculosis are contained in "180111 |
| N. P. 111 . | medical history.xlsx", it should be classified as "with medical history of |
| Medical history: | tuberculosis". When the checkbox of 'medical history unknown' is |
| tuberculosis | checked, it should be 'unknown' while no description should be 'not |
| | provided'. Others are "no medical history of tuberculosis". |
| | When medical-history data on non-tuberculous mycobacteriosis are |
| M. E. 11. | contained in "180111 medical history.xlsx", it should be classified as |
| Medical history: | "with medical history of non-tuberculous mycobacteriosis". When the |
| non-tuberculous | checkbox of 'medical history unknown' is checked, it should be |
| mycobacteriosis | 'unknown' while no description should be 'not provided'. Others are "no |
| | medical history of non-tuberculous mycobacteriosis". |
| | When medical-history data on interstitial pneumonia are contained in |
| | "180111 medical history.xlsx", it should be classified as "with medical |
| Medical history: | history of interstitial pneumonia". When the checkbox of 'medical |
| interstitial pneumonia | history unknown' is checked, it should be 'unknown' while no |
| | description should be 'not provided'. Others are "no medical history of |
| | interstitial pneumonia". |
| | When medical-history data on bronchitis bacterial are contained in |
| Medical history: | "180111 medical history.xlsx", it should be classified as "with medical |
| bronchitis bacterial | history of bronchitis bacterial". When the checkbox of 'medical history |
| | unknown' is checked, it should be 'unknown' while no description |

| Data name | Derivation and calculation methods |
|---|---|
| | should be 'not provided'. Others are "no medical history of bronchitis bacterial". |
| Medical history:<br>aplastic anaemia | When medical-history data on aplastic anaemia are contained in "180111 medical history.xlsx", it should be classified as "with medical history of aplastic anaemia". When the checkbox of 'medical history unknown' is checked, it should be 'unknown' while no description should be 'not provided'. Others are "no medical history of aplastic anaemia". |
| Medical history:<br>pancytopenia | When medical-history data on pancytopenia are contained in "180111 medical history.xlsx", it should be classified as "with medical history of pancytopenia". When the checkbox of 'medical history unknown' is checked, it should be 'unknown' while no description should be 'not provided'. Others are "no medical history of pancytopenia". |
| Medical history:<br>malignant tumour | When medical-history data on malignant tumour are contained in "180111 medical history.xlsx", it should be classified as "with medical history of malignant tumour". When the checkbox of 'medical history unknown' is checked, it should be 'unknown' while no description should be 'not provided'. Others are "no medical history of malignant tumour". |
| Patients with an hepatitis B virus infection | "Hepatitis" "Hepatitis virus carrier" in "Complications" and/or "Medical history" of "1. Patient information" in the survey form → hepatitis viral infections. If "B" in "Complications" and/or "Medical history" is selected, classified the patients as those with hepatitis B virus infection. In addition, a patient with any events of MedDRA PT code provided in "Patients with hepatitis 180111B virus infection.xlsx" should be also classified as a patient with hepatitis B virus infection. |
| Presence/absence of<br>administration of<br>anti-hepatitis B virus<br>agent | If the following drug codes are included in the survey form, regard the case as "with administration of an anti-hepatitis B virus agent". Others are "without administration of an anti-hepatitis B virus agent". Entecavir (Baraclude): 6250029 Tenofovir (Tenozet, Viread): 6250024 Adefovir (Hepsera): 6250026 Lamivudine: 6250006, 6250020 |
| Presence/absence of allergy history | When allergy data are contained in the survey form, it should be classified as "with allergy history". When the checkbox of 'medical history unknown' is checked, it should be 'unknown' while no |

| Data name | Derivation and calculation methods |
|---|---|
| | description should be 'not provided'. Others are "no allergy history". |
| Presence/absence of smoking history | When the checkbox of 'with' smoking history is checked in the survey form, regard it as 'with' smoking history. When the checkbox of 'no' smoking history is checked in the survey form, regard it as 'without' smoking history. When the checkbox of 'unknown' for smoking history is checked in the survey form, regard it as 'unknown'. If nothing is described in the survey form, it should be 'not provided'. |
| Details of smoking<br>history | For the items for smoking history in the survey form, when the 'smoking' checkbox is checked or when the smoking years column is checked of the 'smoking' checkbox, regard it as "smoking". When smoking "in the past" is checked other than "smoking" or when the smoking years for "in the past" is provided, regard it as "only in the past". When a case is not applicable to "smoking" or "only in the past" though a smoking history exists, regard it as "unknown". |
| Administration status | <ul> <li>[1] 1st administration: as a patient with a dose of 160mg</li> <li>[2] 2nd administration: 2nd administration date - the first administration date = 14 days ±4 days or less, and a patient with a dose of 80mg.</li> <li>[3] 3rd administration: 3rd administration date - the 2nd administration date = 14 days ±4 days or less, and a patient with a dose of 40mg.</li> <li>[4] 4th administration and thereafter: the dosing frequency "once every 2 weeks" is checked in the survey form, and a patient with a dose of 40mg <ul> <li>* If the patient receives the fourth administration and thereafter, all the administration status should be the condition as shown in [4].</li> </ul> </li> <li>If all the following [1] to [4] are satisfied, aggregate the data as "160mg→80mg→40mg once every two weeks". Others are aggregated as "others".</li> <li>Of note, when data on administration status include only [1], [2] and [3] or when the data ends halfway for some reason, determine whether the case satisfies the criteria from [1] to [4] as of the final data on</li> </ul> |

| Data name | Derivation and calculation methods |
|---|---|
| | Dosing frequency |
| Administration status<br>(total number of<br>dosing, total dose) | [1] Sort data in the order of "the first administration date" of "the administration status of Humira", dosing frequency and description. [2] Calculate the dosing interval per data on administration status. "When "once every two weeks" is checked, regard it as a 14-day interval. For others, obtain the frequency from "dosing interval". [3] Calculate the dosing frequency per data on administration status. Dosing frequency = (the final administration date (the date imputed based on the definition of 10.1 Final administration date of Humira) — the first administration date(after imputed))/dosing frequency (number of days) When the results of [4] and [3] are ">0" (bigger than 0) and "<1" (smaller than 1), count it as 1. If the figure is ">=1" (1 or bigger), round the decimal down to the integer for the dosing frequency. [5] The total number of dosing shall be the total of [4] per patient. Dose [1] When the dose of Humira is 'others', obtain the dose from "Dose_other description". [2] Calculate the dose per data of the administration status. Dose = the number of dosing * a dose |
| Patients with | <ul> <li>[3] The total dose should be the total of [2] per patient.</li> <li>The mean of a dose</li> <li>The mean of a dose = the total dose/the total number of dosing</li> </ul> |
| self-administration | The patients whose registration form has a check on self-administration. |
| Age | It should be identified based on the date of birth or the first administration date of Humira in the survey form. Of note, if the "date" of birth is incomplete and not provided, impute 1 as the date. When the date of birth is still incomplete even after the above imputation, just mirror the age provided in the survey form. |
| Indication | If multiple checkboxes such as Crohn's disease or others are selected for indication in "1. Patient information" in the survey form, count the number for each indication. Note that Crohn's disease should be selected |

| Data name | Derivation and calculation methods |
|---|---|
| | to display the item of indication in Attachment Form 3. |
| Tuberculin test | Conducted :When the first administration date of Humira is 1 and a day |
| | before the first administration date is -1, the patients who underwent |
| | Tuberculin test between -90 and 1 are regarded as the patients with |
| | Tuberculin test. Of note, the data in the survey form shall be used. |
| | Not conducted: other than the above |
| | Conducted: When the first administration date of Humira is 1 and a day |
| | before the first administration date is -1, the patients who underwent |
| QuantiFeron test | QuantiFeron test between -90 and 1 are regarded as the patients with |
| | QuantiFeron test. Of note, the data in the survey form shall be used. |
| | Not conducted: other than the above |
| | Conducted: When the first administration date of Humira is 1 and a day |
| Name and other was a Mark or proper years | before the first administration date is -1, the patients who underwent |
| Chest X ray test | Chest X ray test between -90 and 1 are regarded as the patients with |
| | Chest X ray test. Of note, the data in the survey form shall be used. |
| | Conducted: When the first administration date of Humira is 1 and a day |
| | before the first administration date is -1, the patients who underwent |
| Thoracic CT test | thoracic CT scan between -90 and 1 are regarded as the patients with |
| | thoracic CT scan. Of note, the data in the survey form shall be used. |
| | Conducted: When the first administration date of Humira is 1 and a day |
| | before the first administration date is -1, the patients who underwent |
| Imaging procedure | chest X ray, thoracic CT scan, or other imaging tests between -90 and 1 |
| | are regarded as the patients with imaging test. Of note, the data in the |
| | survey form shall be used. |
| | The patients who underwent (Tuberculin test or QuantiFeron test) and |
| Tuberculosis test | (chest X ray, thoracic CT scan, or other imaging tests). Of note, the data |
| | in the survey form shall be used. |
| Patients subject to | Patients who are included in "CD Long AAA Measurement (final |
| AAA measurement | report).xlsx". |
| Patients of | The patients whose registration form has at least a check on the |
| contraindications | checkbox of contraindications. |
| Patients who developed | The patients with an infection in an external file "The priority survey |
| an infection | item list_ MedDRA20.1_FIX.xlsx". |
| Patients who developed | The patients with malignant tumour in an external file "The priority |
| malignant tumour | survey item list_MedDRA20.1_FIX.xlsx". |
| Duration of illness (in | "For XX years and XX months" should be converted into the figure in |

| Data name | Derivation and calculation methods |
|---|---|
| years) | years for "duration of illness" of "patient information" in the survey form. When both figures of year and month: year + month/12 When the figure of year is provided: year When the figure of month is provided: month/12 Other cases are identified as "unknown/not provided" as the duration cannot be identified. |
| Concomitant medication | Concomitant medications should the data satisfying the following rules: When concomitant-medication data are contained in the survey form, it should be classified as "with concomitant medications". When "presence/absence of anti-tuberculosis drug", "presence/absence of concomitant medications" in the survey form are not assessable, select "unknown" while they are not provided, select "not provided". Other cases are "without concomitant medications". Data with a drug name in "administration status of anti-tuberculosis drug", "concomitant medications" of the survey form When 'from before Humira administration is started" is checked, the first administration date should be the same as the first administration date of Humira". When the year and month are described for the first administration date of the concomitant medication, impute "1" for the "date". When the year is described for the first administration date of the concomitant medication, impute "1" each for the "month" and "date". When 'continued' is checked, the final administration date should be the same as the final administration date of Humira. When the year and month are described for the final administration date of the concomitant medication, impute the month's final date for the date. When the year is described for the final administration date of the concomitant medication, impute "12" for the month and "31" for the date. When the final administration of concomitant medication < the first administration date of Humira, and/or when the final administration date of Humira < the first administration date of concomitant |

| Data name | Derivation and calculation methods |
|---|---|
| | medication, exclude the case from the calculation for concomitant medication. If the above imputing methods do not help add the date (the first administration date or the final administration date is not provided, etc.), or if the first administration date and the final administration date of concomitant medication are reversed, it should be regarded as a concomitant medication. ('Clear' refers to a condition where no ambiguous expressions like "around", "in the middle", etc. are included and a number or figure only is provided.) |
| Concomitant medication: aminosalicylic acid products | See the drug code list and determine from the drug codes. |
| Concomitant medication: corticosteroid | See the drug code list and determine from the drug codes. |
| Concomitant medication: immunosuppressant | See the drug code list and determine from the drug codes. |
| Concomitant medication: antibiotics | See the drug code list and determine from the drug codes. |
| Concomitant medication: others | Others are the drugs other than aminosalicylic acid products, corticosteroid, immunosuppressant, and antibiotics. |
| Prior medication:<br>TNFα drug | When presence/absence treatment history with anti-TNF $\alpha$ drug is "present" in "treatment history with anti-TNF $\alpha$ drug for Crohn's disease" of the survey form, it should be classified as "with" the history. When the assessment is impossible based on the checkbox, it should be classified as "unknown" whereas no description should be "not provided". Other cases are "without" the history. |
| Prior medications | When a patient had a prior medication of TNFα drug and any of the prior-medication type checkboxes is checked, the patient is regarded as "with prior medications". When the assessment is impossible based on the checkbox of presence/absence of prior medication/treatment, regard it as "unknown" while no description should be "not provided". Other cases are "without" prior medications. |

| Data name | Derivation and calculation methods |
|---|---|
| Prior medication: | If aminosalicylic acid drug in the survey form is checked, regard the |
| aminosalicylic acid | case as "with aminosalicylic acid drug". Others are "without |
| products | aminosalicylic acid drug". |
| Prior medication: | If corticosteroids in the survey form is checked, regard the case as "wit |
| corticosteroid | corticosteroids". Others are "without corticosteroids". |
| Prior medication: | If immunosuppressant in the survey form is checked, regard the case as |
| immunosuppressant | "with immunosuppressant". Others are "without immunosuppressant". |
| Prior medication: | Otherwise, when antibiotics in the survey form is checked, regard the |
| antibiotics | case as "with antibiotics". Others are "without antibiotics". |
| | When any of the checkboxes of each prior-treatment type in "prior |
| | medication/treatment for Crohn's disease is checked in the survey form, |
| Prior treatment | regard it as "with prior treatment". When the assessment is impossible |
| 1 Tior deadliest | based on the checkbox of presence/absence of prior medication/therapy, |
| | regard it as "unknown" while no description should be "not provided". |
| | Other cases are "without" prior treatment. |
| Prior treatment: surgery | Refer to "[Humira CD Long] Conversion data provided for analysis" to |
| 1 Hor treatment, surgery | identify it. |
| Prior treatment: | |
| granulocyte and | When GCAP is checked in the survey form, regard it as "with GCAP". |
| monocyte adsorption | Others are "without GCAP". |
| apheresis (GCAP) | |
| Prior treatment: enteral | When enteral nutrition therapy is checked in the survey form, regard it |
| | as "with enteral nutrition therapy". Others are "without enteral nutrition |
| nutrition therapy | therapy". |
| Prior treatment: | When intravenous nutrition therapy is checked in the survey form, |
| intravenous nutrition | regard it as "with intravenous nutrition therapy". Others are "without |
| therapy | intravenous nutrition therapy". |
| | It should be described in "non-medicinal treatment/concomitant therapy |
| | for Crohn's disease" of the survey form. The data from the first |
| | administration date to the final administration date of Humira will be |
| | calculated. |
| Concomitant therapy | When concomitant-therapy data are contained under the same rule as the |
| | definition of concomitant medications defined in "10.1 General", regard |
| | it "with concomitant therapy". When "presence/absence of concomitant |
| | therapy" in the survey form is not assessable, select "unknown" while it |
| | is not provided, select "not provided". Other cases are "without |

| Data name | Derivation and calculation methods |
|---|---|
| | concomitant therapy". |
| Concomitant therapy: surgery | Refer to "[Humira CD Long] Conversion data provided for analysis" to identify it. |
| Concomitant therapy:<br>GCAP | When GCAP is checked in the survey form, regard it as "with GCAP". Others are "without GCAP". |
| Concomitant therapy:<br>enteral nutrition<br>therapy | When enteral nutrition therapy is checked in the survey form, regard it as "with enteral nutrition therapy". Others are "without enteral nutrition therapy". |
| Concomitant therapy:<br>intravenous nutrition<br>therapy | When intravenous nutrition therapy is checked in the survey form, regard it as "with intravenous nutrition therapy". Others are "without intravenous nutrition therapy". |
| Work condition | Just mirror the checked information at "work condition" in the survey form. Of note, if multiple checkboxes are checked or the check is not assessable, regard it as "unknown". When none of the items are checked, it should be "not provided". |

## 10.2. Safety analysis

| Data name | Derivation and calculation methods |
|---|---|
| | The adverse events for analysis should include not only the events |
| | derived from the survey form but also the events covered in the detailed |
| | investigation which has been described by the physicians at a contracted |
| | site/department even though not derived from the survey form in |
| | "Humira CD Long_AE matching list". |
| Adverse event | With adverse event: at least 1 record on adverse event(s) exists |
| | Without adverse event: other than the above. |
| | When adverse events are counted per SOC, the identical SOC in a |
| | patient should be counted as 1 whereas the same PT in the same patient |
| | be counted as 1 for PT. When no applicable patients were observed, |
| | display "0" for the number of patients and "0.00" for the percentage. |
| | Based on the seriousness criteria for company assessment which are |
| | provided in "Humira CD Long_AE matching list", regard the events |
| Caniana and a factoria | which have been assessed to be serious as serious adverse events. |
| Seriousness of adverse<br>events | With serious adverse event: at least 1 record on serious adverse event(s) |
| | exists |
| | Without serious adverse event: other than the above. |
| | Follow the way of counting adverse events to count serious adverse |

| Data name | Derivation and calculation methods |
|---|---|
| | events. |
| | Give the following priority to serious adverse events for aggregation. |
| | [1]serious [2]non-serious |
| | Unless a serious adverse event is assessed as "not related" in the |
| Coursel relationship of | company causality assessment provided in "Humira CD Long_AE |
| Causal relationship of adverse events | matching list", regard the event as 'with' causal relationship. Give the |
| adverse events | following priority to causal relationship for aggregation. |
| | [1] With causal relationship [2] without causal relationship |
| | Use the outcomes for company assessment provided in "Humira CD |
| | Long_AE matching list" to give the following priority to the outcomes |
| Outcome of adverse | for aggregation based on the rules in "derivation and calculation |
| events | methods" for adverse events. |
| | [1] [1] death [2] unknown [3] not recovered [4] recovered with sequela |
| | [5] recovering [6] recovered [7] not provided |
| | Use the onset date for company assessment provided in "Humira CD |
| | long-term_AE matching list". |
| | When the first administration date of Humira and the adverse-event |
| | onset date can be identified as the complete date, they can be used for |
| Days from the first | calculation. |
| administration date of | When the first administration date of Humira <= the adverse-event onset |
| Humira to the | date: |
| adverse-event onset | Adverse-event onset date - the first administration date of Humira + 1 |
| date | When the first administration date of Humira > the adverse-event onset |
| | date: |
| | Adverse-event onset date - the first administration date of Humira |
| | When more than one identical PT is found in a patient, use the first |
| | onset date to identify the adverse event to be counted. |
| | Use the onset date and the outcomes (recovered or recovering) for |
| Days from the | company assessment provided in "Humira CD Long_AE matching list". |
| adverse-event onset | When the adverse-event onset date and the outcome confirmation date |
| date to the outcome | can be identified as the complete date, they can be used for calculation. |
| confirmation date | Outcome confirmation date - adverse-event onset date + 1 |
| (recovered or | When more than one identical PT is found in a patient, choose the event |
| recovering) | which persisted longest until the recovery or the outcome confirmation |
| | date. |

| Data name | Derivation and calculation methods |
|---|---|
| Incidence of adverse | Calculate the incidence of adverse reactions, incidence of serious |
| reactions, incidence of | adverse reactions, incidence of adverse events, incidence of serious |
| serious adverse | adverse events with the number of patients with any of the |
| reactions, incidence of | reactions/events in numerator and the number of patients in the safety |
| adverse events, | analysis group in denominator. |
| incidence of serious | Provide how to calculate in each table at Chapter 13 and thereafter if |
| adverse events | other calculation methods are used. |

## 10.3. Effectiveness analysis

| Data name | | Derivation and calculation method | s |
|---|---|---|---|
| Remission | When the | When the CDAI score is <150, the case is regarded as remission. | |
| | Q1 | Do you work now? | Yes, no |
| | Q2 | How many hours did you leave the work due to problems related to Crohn's disease over the past 7 days? | () hour(s) |
| | Q3 | How many hours did you leave the work<br>for a reason other than Crohn's disease<br>such as holidays or hours for which you<br>were off to participate in this survey<br>over the past 7 days? | () hour(s) |
| | Q4 | How many hours did you actually work for the past 7 days? | () hour(s) |
| WPAI | Q5 | How much productivity was affected by Crohn's disease while you were working over the past 7 days? 0: Crohn's disease did not affect the work. 10: Crohn's disease completely interrupted the work. Based on the above, your score between 0 to 10. | ( ) |
| | Q6 | How much did Crohn's disease affect various daily activities except your job over the past 7 days? | ( ) |

| Data name | Derivation and calculation methods |
|---|---|
| | 0: Crohn's disease did not affect daily activities. 10: Crohn's disease completely interrupted daily activities. Based on the above, your score between 0 to 10. |
| | • Absenteeism (%) Calculate it with the following formula based on the questions (Q1 to Q6) on the above table: [Q2/(Q2+Q4)] × 100 |
| | <ul> <li>Presenteeism (%)</li> <li>Calculate it with the following formula based on the questions (Q1 to Q6) on the above table:</li> <li>(Q5 / 10) × 100</li> </ul> |
| | <ul> <li>Overall work impairment (%) Calculate it with the following formula based on the questions (Q1 to Q6) on the above table: {Q2/(Q2+Q4)+[1-Q2/(Q2+Q4)]×(Q5/10)} × 100 </li> <li>Activity Impairment (%) Calculate it with the following formula based on the questions (Q1 to </li> </ul> |
| | Q6) on the above table: $(Q6/10) \times 100$ |

## 11. How to stratify data

| Data | How to stratify |
|---|---|
| Dosage and | 160mg→80mg→40mg once every two weeks, other |
| administration | 100mg—80mg—40mg once every two weeks, other |
| | ≥1 and <4, |
| | ≥4 and <13, |
| | ≥13 and <26, |
| Dosing frequency | ≥26 and <39, |
| (times) | ≥39 and <52, |
| | ≥52 and <65, |
| | ≥65 and <78, |
| | ≥78 |
| | <500mg, |
| | ≥500mg and <1000mg |
| Total days (mas) | ≥1000mg and <2000mg |
| Total dose (mg) | ≥2000mg and <3000mg |
| | ≥3000mg, |
| | Unknown |
| | the first administration to Week 4 of administration, |
| | after Week 4 of administration to Month 3 of administration, |
| | after Month 3 of administration to Month 6 of administration, |
| | after Month 6 of administration to Year 1 of administration, |
| Dose period | after Year 1 of administration to Year 1 and Month 6 of administration, |
| | after Year 1 and Month 6 of administration to Year 2 of administration, |
| | after Year 2 of administration to Year 2 and Month 6 of administration, |
| | after Year 2 and Month 6 of administration to Year 3 of administration, |
| | Continued as of Year 3 of administration |
| Reason for | Development of adverse event, lack of effectiveness, patient's wish, no |
| discontinuation | visit, others |
| Sex | Man, women, unknown/not provided |
| Pregnancy/nursing | Not pregnant/nursing, pregnant, nursing, unknown/not provided |
| Age (in years) | <15, ≥15 and <65, ≥65, unknown/not provided |
| Dodowaiał (I-) | <30, ≥30 and <40, ≥40 and <50, ≥50 and <60, ≥60, unknown/not |
| Body weight (kg) | provided |
| BMI(kg/m <sup>2</sup> ) | <18.5, ≥18.5 and <25, ≥25 and <30, ≥30, unknown |
| Duration of illness (in | <2, ≥2 and <5, ≥5 and <10, ≥10, unknown/not provided |

| Data | How to stratify |
|---|---|
| years) | |
| Indication | Crohn's disease, other, unknown/not provided |
| Allergy history | Without the history, with the history, unknown/not provided |
| Smoking history | Without the history, with the history, unknown/not provided |
| Details of smoking history | Smoking, only in the past (not smoking now), unknown |
| HBs antigen | Not conducted, conducted, unknown/not provided |
| Tuberculosis-test status | Not conducted, conducted |
| Complications | Without the history, with the history, unknown/not provided |
| Detailed classification of complications | Liver disorder, renal disorder, blood disorder, respiratory disorder, others |
| Other classification of complications | Diabetes mellitus, osteoporosis, malignant tumour, others |
| Medical history | Without the history, with the history, unknown/not provided |
| Detailed classification of medical history | Tuberculosis, non-tuberculous mycobacteriosis, interstitial pneumonia, bronchitis bacterial, aplastic anaemia, pancytopenia, malignant tumour, others |
| Prior medications for<br>Crohn's disease | Without the history, with the history, unknown/not provided |
| Detailed classification<br>of prior medications for<br>Crohn's disease | Anti-TNF $\alpha$ drug, aminosalicylic acid products, corticosteroid, immunosuppressant, and antibiotics. |
| Prior treatment for<br>Crohn's disease | Without the history, with the history, unknown/not provided |
| Detailed classification<br>of prior treatment for<br>Crohn's disease | Surgery, GCAP, enteral nutrition therapy, intravenous nutrition therapy, others |
| Treatment history with anti-TNFα drug | Without the history, with the history, unknown/not provided |
| Reason for<br>discontinuation of<br>treatment history with<br>anti-TNFα drug | Lack of efficacy, adverse events, others, unknown/not provided |
| Concomitant medication | Without the history, with the history, unknown/not provided |
| Detailed classification | Aminosalicylic acid products, corticosteroid, immunosuppressant, |

| Data | How to stratify |
|---|---|
| of concomitant | antibiotics, and others |
| medications | |
| Concomitant therapy | Wat of the state o |
| for Crohn's disease | Without the history, with the history, unknown/not provided |
| Detailed classification | c com a large d |
| of concomitant therapy | Surgery, GCAP, enteral nutrition therapy, intravenous nutrition therapy, |
| for Crohn's disease | others |
| Condition/site of | |
| disease in the medical | Anus/perianal region, rectum, stomach/duodenum, colon, jejunum/ileum, |
| history of Crohn's | other, unknown/not provided |
| disease | |
| Intestinal complications | |
| as condition/site of | |
| disease in the medical | Without the history, with the history, unknown/not provided |
| history of Crohn's | |
| disease | |
| Non-intestinal | |
| complications as | |
| condition/site of | |
| disease in the medical | Without the history, with the history, unknown/not provided |
| history of Crohn's | |
| disease | |
| | Routinely engaged in wage labor for 35 hours or longer a week, |
| | Routinely engaged in wage labor for 35 hours or less a week, |
| | Not engaged in wage labor but do housework, shopping, childrearing, |
| Work condition | exercise, or study |
| | , Involved in daily living activities, |
| | Involved in less daily activities due to hospitalization, etc. |
| | Unknown/not provided |
| | <150: remission |
| CDAI at the fact | ≥150 and <220: mild |
| CDAI at the first administration | ≥220 and <450: moderate |
| | >450: severe |
| | Unknown/not provided |
| CDD | <1.0mg/dL, |
| CRP | ≥1.0mg/dL, |

| Data | How to stratify |
|---|---|
| | Unknown/not provided |
| Self administration | Without the history, with the history, unknown/not provided |

## 12. Data handling at test/assessment periods

## 12.1. Assessment period for CDAI, WPAI, CRP and non-intestinal conditions

Time allowance of assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Time Allowance(Day) |
|---|---|
| At the first administration | - 1 (scheduled date 1) |
| Week 4 of administration | 15 - 43 (scheduled date 29) |
| Month 3 of administration | 71 - 99 (scheduled date 85) |
| Month 6 of administration | 169 - 197 (scheduled date 183) |
| Year 1 of administration | 337 - 393 (scheduled date 365) |
| Year 1 and Month 6 of administration | 519 - 575 (scheduled date 547) |
| Year 2 of administration | 701 - 757 (scheduled date 729) |
| Year 2 and Month 6 of administration | 883 - 939 (scheduled date 911) |
| Year 3 of administration | 1065 - 1121 (scheduled date 1093) |
| At final assessment | Final assessment of each patient no matter whether the each assessment period is within Time Allowance. |

The data for analysis should derive from the date closest to the scheduled date within Time Allowance. If there are more than one data dated on the same day, select the worst value.

## 12.2. Assessment period of endoscopy results

Time allowance of assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Time Allowance(Day) |
|---|---|
| At the first administration | - 1 (scheduled date 1) |
| Month 6 of administration | 2 - 182 (scheduled date 183) |
| Year 1 of administration | 183 - 364 (scheduled date 365) |
| Year 2 of administration | 365 - 728 (scheduled date 729) |
| Year 3 of administration | 729 - 1092 (scheduled date 1093) |
| At final assessment | Final assessment of each patient no matter whether the each assessment period is within Time Allowance. |

The data for analysis should derive from the date closest to the scheduled date within Time Allowance. If there are more than one data dated on the same day, select the worst value.

## 12.3. Assessment period for the administration status of Humira

Time allowance of assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Time Allowance(Day) |
|---|---|
| the first administration to Week 4 of administration | 1-28 |
| after Week 4 of administration to Month 3 of administration | 29-84 |
| after Month 3 of administration to Month 6 of administration | 85-182 |
| after Month 6 of administration to Year 1 of administration | 183-364 |
| after Year 1 of administration to Year 1 and<br>Month 6 of administration | 365-546 |
| after Year 1 and Month 6 of administration to<br>Year 2 of administration | 547-728 |
| after Year 2 of administration to Year 2 and<br>Month 6 of administration | 729-910 |
| after Year 2 and Month 6 of administration to<br>Year 3 of administration | 911-1092 |
| Continued as of Year 3 of administration | 1093-, patients with 'continued' checked |

## 12.4. Assessment period for the onset status of adverse reactions

Time allowance of assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Time Allowance(Day) |
|---|---|
| the first administration to Week 4 of administration | 1-28 |
| after Week 4 of administration to Month 3 of administration | 29-84 |
| after Month 3 of administration to Month 6 of administration | 85-182 |
| after Month 6 of administration to Year 1 of administration | 183-364 |
| after Year 1 of administration to Year 1 and<br>Month 6 of administration | 365-546 |
| after Year 1 and Month 6 of administration to<br>Year 2 of administration | 547-728 |
| Assessment period | Time Allowance(Day) |
|---|---|
| after Year 2 of administration to Year 2 and<br>Month 6 of administration | 729-910 |
| after Year 2 and Month 6 of administration to<br>Year 3 of administration | 911-1092 |
| Year 3 of administration - | 1093 - |

## 12.5. Assessment period for the continued administration of Humira

The assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Day |
|--------------------------------------|------|
| At the first administration | 1 |
| Week 4 of administration | 29 |
| Month 3 of administration | 85 |
| Month 6 of administration | 183 |
| Year 1 of administration | 365 |
| Year 1 and Month 6 of administration | 547 |
| Year 2 of administration | 729 |
| Year 2 and Month 6 of administration | 911 |
| Year 3 of administration | 1093 |

# 13. Charts to be generated (chart No., chart name)

#### 13.1. General

## "1.1.1 Case structure chart"

Patients for analysis: registered patients

Analysis objective: to indicate changes in the number of patients

Analysis items: number of sites with registered patients, number of registered patients, number of sites with patients whose survey form has been locked, number of patients whose survey form was locked, number of patients whose survey form was yet to be locked, the breakdown of the reasons for unlocked survey forms, number of patients in the safety analysis group, number of patients excluded from the safety analysis group, the breakdown of reasons for exclusion from the safety analysis group, number of patients in the effectiveness analysis group, number of patients excluded from the effectiveness analysis group, the breakdown of reasons for exclusion from the effectiveness analysis group

"1.1.2 Case structure chart on patients in the effectiveness analysis group" Patients for analysis: patients in the effectiveness analysis group Analysis objective: to indicate changes in the number of patients

Analysis items: number of patients in the effectiveness analysis group, number of patients in the CRP analysis group, number of patients in the WPAI analysis group, number of patients in the endoscopy (large intestine) analysis group, and number of patients in the endoscopy (small intestine) analysis group

Note: the definitions of patients in each analysis group are as follows:

Patients in the CRP analysis group: the patients in the effectiveness analysis group whose CRP level was measured after they were started on Humira.

Patients in the WPAI analysis group: the patients in the effectiveness analysis group whose WPAI was measured after they were started on Humira.

Patients in the endoscopy (large intestine) analysis group: the patients in the effectiveness analysis group who underwent endoscopy (large intestine) after they were started on Humira.

Patients in the endoscopy (small intestine) analysis group: the patients in the effectiveness analysis group who underwent endoscopy (small intestine) after they were started on Humira.

"1.2 Number of sites surveyed and number of patients surveyed (patients in the safety analysis group)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the number of patients per site

Analysis items: number of sites surveyed, number of patients in the safety analysis group, the mean, the maximum, the minimum of the number of patients in the safety analysis group per site

## "1.1.3 Progress in survey forms"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show the number of locked cases for each separate volume per patients whose survey form was locked, patients in the safety analysis group, and patients in the effectiveness analysis group.

Analysis items: locked cases in the 1st separate volume, locked cases in the 2nd separate volume, locked cases in the 3rd separate volume, locked cases in the 4th separate volume, locked cases in the 5th separate volume, locked cases in the 6th separate volume

"1.3 A list of the patients excluded from the safety analysis and the patients excluded from the effectiveness analysis (including the reason for exclusion)"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show the list of patients excluded from each analysis group and the reason for exclusion

Analysis item: The reason for exclusion will be displayed for the patients not in the safety or efficacy

analysis.

If more than one reason for exclusion exists in a patient, display them in a comma-delimited manner.

#### "1.3.1. Excluded patients (aggregation by reason)"

Patients for analysis: registered patients

Analysis objective: to show a list of the reasons for exclusion in each analysis group regarding all the patients in the analysis group.

Analysis items: case number, patients whose survey form was yet to be locked, patients excluded from the safety analysis group, the reasons for exclusion from the safety analysis (breach of contract: unsigned site/department, breach of contract: unsigned physician, breach of contract: an excess of the number of signed patients, untreated with Humira, administration prior to contract, administration after the contract expires, administration start not in the registration period, breach of registration criteria: deviation of the registration period, breach of registration criteria: not the disease surveyed, breach of registration criteria: malignant tumour, breach of registration criteria: during the administration period of Humira, not confirmed by physician, patients not registered, overlapped patients, safety not assessable, data credibility not confirmed, data credibility not confirmed (breakdown)), patients excluded from the effectiveness analysis, reasons for exclusion from the effectiveness analysis (effectiveness not assessable)

If data credibility cannot be identified and more than one (breakdown) exists in a patient, display them in a comma-delimited manner.

#### "1.4 A list of patients (adverse event + search flag)"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of background information per patient, adverse events and administration status by using analysis data.

Analysis items: case number, sex, age, body weight, duration of illness, adverse event (presence/absence of adverse event, safety

Patients with adverse events not in the analysis period, SOC code, System Organ Class, PT code, name of disease (MedDRA PT), adverse events reported by physician, onset date, days from the first administration to the onset, seriousness, causality, outcome, outcome confirmation date, days to the outcome confirmation), CDAI effectiveness at the final assessment, administration status of Humira (the first administration date, the final administration date, days of administration, the initial dose, the maximum dose) presence/absence of complication, presence/absence of medical history, hepatitis B virus test (HBs antigen), with/without administration of anti-hepatitis B virus agent, tuberculosis test (Tuberculin test, QuantiFeron test, chest X ray test, thoracic CT scan, other imaging, tuberculosis test) search flags (patients in the safety analysis group, patients in the effectiveness analysis group, death cases, pediatrics, the elderly, pregnant, nursing, liver disorder, renal disorder, patients with hepatitis B viral infection, patients with an infection, patients with malignant tumour,

patients with AAA measured, contraindication)

Note: Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for CDAI effectiveness in the final assessment period.

In addition, display "remission" or "no remission". Display "unknown" for patients excluded from the effectiveness analysis.

#### "1.4.1 A list of adverse events"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of adverse events per patient by using analysis data.

Analysis items: case number, sex, age, SOC code, System Organ Class, PT code, name of disease (MedDRA PT), adverse events reported by physician, onset date, days from the first administration date to the onset date, seriousness, causality,

outcome, outcome confirmation date, dates to the outcome, complication, patients in the safety analysis group, the reasons for exclusion from the safety analysis (breach of contract: unsigned site/department, breach of contract: unsigned physician, breach of contract: an excess of the number of signed patients, untreated with Humira, administration prior to contract, administration after the contract expires, administration start not in the registration period, breach of registration criteria: deviation of the registration period, breach of registration criteria:

not the disease surveyed, breach of registration criteria: malignant tumour, breach of registration criteria: during the administration period of Humira, not confirmed by physician, patients not registered, overlapped patients, safety not assessable, data credibility not confirmed, data credibility not confirmed (breakdown)), patients in the effectiveness analysis group, patients who developed adverse events not in the safety analysis period, search flag (death case, pediatrics, the elderly, pregnant, nursing, liver disorder, renal disorder, patients with hepatitis B viral infection, patients with an infection, patients with malignant tumour, patients with AAA measured, contraindication)

If data credibility cannot be identified and more than one (breakdown) exists in a patient, display them in a comma-delimited manner.

## "1.4.2 A list of death cases"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of adverse events in death cases by using analysis data.

Analysis items: case number, sex, age, SOC code, System Organ Class, PT code, name of disease (MedDRA PT), adverse events reported by physician, onset date, days from the first administration date to the onset date, seriousness, causality,

outcome, outcome confirmation date, days to the outcome, complication, patients in the safety analysis group, patients in the effectiveness analysis group, patients who developed adverse events not in the safety analysis period, search flag (death case, pediatrics, the elderly, pregnant, nursing,

liver disorder, renal disorder, patients with hepatitis B viral infection, patients with an infection, patients with malignant tumour, patients with AAA measured, contraindication)

# "1.4.3 A list of patients aged 18 years or younger"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of patients aged 18 years or younger by using analysis data.

Analysis items: case number, sex, age, height, body weight, BMI, duration of illness, adverse event (SOC code, System Organ Class, PT code, name of disease (MedDRA PT), adverse events reported by physician, onset date, days from the first administration date to the onset date, seriousness, causality, outcome, outcome confirmation date, days to the outcome), administration status of Humira (the first administration date, the final administration date), discontinued/not discontinued, reason for discontinuation, complication (presence/absence of complication, PT code, name of disease (MedDRA PT), medical history (presence/absence of medical history, PT code, name of disease (MedDRA PT)), condition/ medical history of Crohn's disease (anus/perianal region, rectum, stomach/duodenum, colon, jejunum/ileum, others, intestinal complication, non-intestinal complication), prior medications (anti-TNFα drug, aminosalicylic acid drug, corticosteroids, immunosuppressant, antibiotics), CDAI level (at the first administration, Week 4 of administration, Month 3 of administration, Month 6 of administration, Year 1 of administration, Year 1 and Month 6 of administration, Year 2 of administration, Year 2 and Month 6 of administration , Year 3 of administration)

Note: Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for CDAI level.

## "1.5 Administration status of Humira (dosage and administration)"

Patients for analysis: patients in the safety analysis group, patients in the effectiveness analysis group

Analysis objective: to show the administration status of Humira

Analysis items: count the number of patients who receive Humira in the process of "1st time:  $160 \text{mg} \rightarrow 2 \text{nd}$  time:  $80 \text{mg} \rightarrow 3 \text{rd}$  time: 40 mg once every two weeks, and no change thereafter" and the number of "other" patients, and calculate the percentage to the target patients. See 10.1 for how to classify the administration process.

# "1.6.1 Administration status of Humira (dosing frequency, dose)

Patients for analysis: patients in the safety analysis group, patients in the effectiveness analysis group

Analysis objective: to show the dosing frequency and the distribution status of the total dose Analysis items: calculate the number of patients per segment defined in "11 How to stratify data", summary statistics and the percentage to the number of patients in the analysis groups regarding dosing frequency and the total dose.

#### "1.6.2 Administration status of Humira (period)"

Patients for analysis: patients in the safety analysis group, patients in the effectiveness analysis group

Analysis objective: to show the distribution status in the administration period.

Analysis item: Calculate the administration dates based on "days to the final administration date of Humira" of "10.1 General" for the administration period. Then, calculate the number of patients per segment which contains the administration dates in each patient and the percentage to the patients in the analysis group in the Time Allowance defined in "12.3 Assessment period for administration status of Humira". In addition, calculate summary statistics for the number of days for administration.

## "1.6.3 Continuation rate of Humira"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the continuation rate of Humira using the Kaplan-Meier method.

Analysis items: Calculate At Risk, number of discontinued patients, continuation rate and 95% of continuation rate per assessment period.

Generate the Kaplan-Meier curve with the percentage of the number of discontinued patients to At Risk as the continuation rate.

Note: Follow "12.5 Assessment period for the continuation of Humira administration" for the dates of assessment period.

The days are censored at the first administration date of Humira + 1092 in patients who are still registered at Year 3.

Calculate the analysis items using the Kaplan-Meier method.

At Risk should include the number of patients who are exposed to a discontinuation risk.

## "1.7 Administration status of Humira (discontinuation of administration)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the number of discontinued patients and the breakdown of the reasons for discontinuation.

Analysis items: Calculate the number of patients in the analysis groups, the percentage to the discontinued patients and patients in the analysis groups, patients 'with' reason for discontinuation and unknown/not provided and the percentage to the number of discontinued patients, number of patients per "reason for discontinuation" defined in "11 How to stratify data" and the percentage to the number of discontinued patients.

Note: the reasons for discontinuation may be overlapped in calculation.

In addition, if there are no patients applicable to "multiple choices", do not display the items of "multiple choices".

# "1.7.1 Administration status of Humira (reason for discontinuation other reasons)

Patients for analysis: patients in the safety analysis group

Analysis objective: to show a list in which the reason for discontinuation is 'others'.

Analysis item: Calculate the number of patients classified into "others "of "reasons for discontinuation" defined in "11 How to stratify data" by classified item of "reasons for discontinuation, other reason".

# "1.7.2 Administration status of Humira (a list of reasons for discontinuation other reasons)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show a list in which the reason for discontinuation is 'others'.

Analysis item: Display other reasons per case number for patients classified into "others" of "reasons for discontinuation" defined in "11 How to stratify data".

# "1.12 Distribution status of patient backgrounds"

Patients for analysis: patients in the safety analysis group, patients in the effectiveness analysis group, patients whose survey form was locked

Analysis objective: to show the distribution status of patient backgrounds

Analysis item: calculate the number of patients in the analysis groups.

Calculate the number of patients per the following segment defined in "11 How to stratify data" and the percentage to the number of patients in the analysis groups.

Sex, pregnancy/nursing, age (year), body weight (kg), BMI (kg/m²), duration of illness (year), indication (registration form), allergy history, smoking history, detailed classification of smoking history, tuberculosis test, hepatitis B virus test status (registration form), complication, detailed classification of complications, complication/others, medical history, detailed classification of medical history, prior medication for Crohn's disease, detailed classification of prior medication for Crohn's disease, prior treatment for Crohn's disease, detailed classification of prior treatment for Crohn's disease, treatment history with anti-TNFα drug for Crohn's disease, reason for discontinuation of treatment history of anti-TNFα drug, concomitant medication, detailed classification of concomitant medications, concomitant treatment for Crohn's disease, detailed classification of concomitant treatment for Crohn's disease, condition/medical history of Crohn's disease (site of disease of condition/medical history of Crohn's disease), intestinal complications of condition/medical history of Crohn's disease, non- intestinal complications of condition/medical history of Crohn's disease), work condition, CDAI when the administration was started, CRP In addition, calculate summary statistics for the following:

age (year), body weight (kg), BMI (kg/m<sup>2</sup>), duration of illness (year), CDAI when the administration was started, CRP

Note: for pregnancy/nursing, calculate the percentage to female patients.

Note: For the discontinuation reasons for anti-TNF $\alpha$  drug, calculate the percentage to the patients with treatment history of anti-TNF $\alpha$  drug.

## "1.13 Distribution status of self-administration"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the distribution status regarding presence/absence of self-administration Analysis item: calculate the number of patients in the analysis groups.

Calculate the number of patients per "self-administration" defined in "11. How to stratify data" and the percentage to the number of patients in the analysis groups.

# "1.16 A list of patients with AAA measured

Patients for analysis: patients in the safety analysis group

Analysis objective: to show a list of patients with AAA measured.

Analysis item: display the following items in "patients with AAA measured" defined in "10.1 General".

Case number, administration status of Humira (the first and final administration dates), concomitant medications, serum anti-adalimumab antibody (blood sampling date, positive/negative) adverse events reported by physician, name of disease (MedDRA PT), System Organ Class, onset date, seriousness, causality, outcome confirmation date, outcome, CDAI remission

# 13.2. Safety

"2.2 A list of the onset status of serious adverse events (Attachment Form 10)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of serious adverse events

Analysis item: aggregate the following items per period for adverse events which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of sites surveyed, number of patients surveyed, number of patients with serious adverse events, number of serious adverse events, incidence of adverse events, incidence of serious adverse events and type of adverse reactions, etc. (SOC, PT).

Note: The classification of period should include at approval, cumulative and total.

Put \* before the PT of unexpected events from "Precautions".

"2.3 A list of target-patient summary (Attachment Form 3)"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of patients

Analysis item: provide the items for analysis and the definitions below.

(1) Case number

Provide a serial number starting 1 per patient.

(2) Name of site (company code)

Describe it in Japanese, as the official name. Obtain the name of site from "[CD Long-term]DCF code list\_Company A.xlsx" and "[CD Long-term]DCF code list\_Company E.xlsx".

(3) Main establishing entity/code

Obtain the code from "Ultmarc re-examination classification".

(4) Name of prefecture where the business is located

Fill in the name. Obtain the prefecture's name from "Ultmarc re-examination classification 2015 0731.xlsx".

(5) Patient abbreviation name

Fill in "not applicable" as mentioned in GB.

(6) Sex

Fill in man, women, unknown or not provided as mentioned in GB.

(7) Date of birth (or age)

Unify it in age. Fill in "A + age + "0000" as mentioned in GB.

(8) Inpatient/outpatient

Fill in inpatient, outpatient, unknown or not provided as mentioned in GB.

(9) Indication

Code, name of disease: Obtain the MedDRA/J LLT code and LLT from the indication of Humira described in the survey form.

(10) Severity prior to administration

Note: Follow Time Allowance of "12.1 Assessment period for CDAI, WPAI, CRP to show CDAI when the administration was started at the following 4 levels:

<150: remission, ≥150 and <220: mild, ≥220 and ≤450: moderate, >450: severe in severity

# (11) Complications

Presence/absence: Refer to the "presence/absence of complications" defined in "10.1 General".

Number of described complications: the number of PT codes encoded by MedDRA/J. If more than 1 identical PT code is found in a patient, count the PT as 1. Describe "0" for the case with no complications.

Term: Describe the PT of complication encoded by MedDRA/J. Arrange detailed classification of complication, the name of complication disease name, a serial number of the complication per patient. Leave the column blank for the case with no descriptions.

#### (12) Route of administration

Describe it as "SC".

#### (13) Maximal dose (a dose)

The maximum of a dose Select the largest number in "administration status defined in "10.1 General" per patient.

#### (14) The mean dose (a dose)

The mean of a dose

It should be the value of "total dose/total dosing times" based on the "administration status (total dosing time, total dose)" defined in "10.1 General".

## (15) Unit

Use "MG".

# (16) daily dosing frequency (the maximum)

Use "1".

# (17) Period for administration

The value of "total dosing time" based on "administration status (total dosing time, total dose)" defined in "10.1 General".

# (18) Concomitant medications

Drug code, the principal drug name: arrange concomitant medications for Crohn's disease (the concomitant medications checked at the indication: Crohn's disease in the survey form) per patient in the order of separate volume and description, and choose the concomitant medication data at the top. If there is no concomitant medication, leave the drug code column blank, and the name of the primary drug "null".

Number of descriptions: count the number of the drug codes for concomitant medications arranged with the rule mentioned above. If more than 1 identical drug code is found in a patient, count it as 1 (for all the concomitant medications no matter whether the indication: Crohn's disease is checked). Describe "0" for the case with no concomitant medications.

# (19) Effectiveness level

Follow Time Allowance of "12.1 Assessment period for CDAI, WPAI, CRP and no-intestinal conditions" to display remission/non-remission at the final assessment. Of note, if remission/non-remission at the final assessment is not reported, regard it as "unknown".

# (20) Adverse reactions

Handle the events with the identical PT code in a patient as 1 record regarding adverse events which occurred in the safety analysis period.

Organ-name code: select the SOC code. When presence/absence is "absence", leave the column blank.

Adverse reaction code: select the PT code. When presence/absence is "absence", leave the column blank.

Name of adverse reactions: select the PT. When presence/absence is "absence", leave the column

blank.

Presence/absence: Select "present" for the data with both adverse events and causal relationship among the adverse reactions which occurred in the safety analysis period. If presence/absence of adverse events is unknown, select "unknown". If presence/absence of adverse events is not provided, select "not provided". Others are "absent". If the reason is 'safety assessment cannot be made' in the patients excluded from the safety analysis, select "unknown".

Number of descriptions: count the number of PT codes. If more than 1 identical PT code is found in a patient, count the PT as 1.

When presence/absence is "absence", leave the column blank.

#### (21) Outcome

For PT codes displayed for adverse reactions, select the outcome with the highest priority in the "outcome" priorities defined in "10.2 Safety analysis". When presence/absence of adverse reactions is "absence", leave the column blank.

# (22) Survey form number

Use the case number in this study.

#### (23) Dropout

If a patient is dropped out from both the safety analysis and the effectiveness analysis, display the case as "both dropout".

If a patient is dropped out only from the safety analysis, display the case as "Safe dropout".

"If a patient is dropped out only from the effective analysis, display the case as "Effective\_dropout".

Note: If there are no applicable data in an aggregation column, display "0" and no columns should be left blank.

# "2.4.1.1 A list of the onset status of adverse reactions (priority survey items)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the summary statistics on the days to the onset as well as the number of patients per outcome and the days to the confirmed outcome (recovered or recovering) for adverse reactions of the priority survey items.

Analysis items: calculate the number of cases and the percentage to the number of patients in the analysis groups per type of adverse reactions (priority survey item, PT), and the number of patients with serious reactions and the percentage to the number of patients in the analysis groups regarding the adverse reactions which occurred in the safety analysis period. In addition, calculate the summary statistics (the number of patients, the mean, the minimum, the median, the maximum) for days to the onset per PT and priority survey item (for the total number of PTs) and for days from the onset date to the outcome (recovered or recovering) as well as the number of patients per outcome.

Note: When more than one identical PT is found in a patient, aggregate seriousness, days to the onset, outcome and days to the outcome (recovered or recovering) as 1 patient (case) in the following manner.

- Seriousness priority: serious > non-serious
- Days to the onset: identify the days as mentioned in "10.2 days from the first administration date of Humira to the adverse-event onset date".
- Outcome: identify it as mentioned in "10.2 Outcome".
- Days to outcome (recovered or recovering): identify the days as mentioned in 10.2 Days from an onset date of adverse events to the outcome confirmation date (recovered or recovering).

# "2.4.1.2 A list of the onset status of adverse events (priority survey items)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the summary statistics on the days to the onset as well as the number of patients per outcome and the days to the confirmed outcome (recovered or recovering) for adverse events of the priority survey items.

Analysis items: calculate the number of cases and the percentage to the number of patients in the analysis groups per type of adverse events (priority survey item, PT), and the number of patients with serious events and the percentage to the number of patients in the analysis groups regarding the adverse events which occurred in the safety analysis period. In addition, calculate the summary statistics (the number of patients, the mean, the minimum, the median, the maximum) for days to the onset per PT and priority survey item (for the total number of PTs) and for days from the onset date to the outcome (recovered or recovering) as well as the number of patients per outcome.

Note: When more than one identical PT is found in a patient, aggregate seriousness, days to the onset, outcome and days to the outcome (recovered or recovering) as 1 patient (case) in the following manner.

- Seriousness priority: serious > non-serious
- Days to the onset: identify the days as mentioned in "10.2 days from the first administration date of Humira to the adverse-event onset date".
- Outcome: identify it as mentioned in "10.2 Outcome".
- Days to outcome (recovered or recovering): identify the days as mentioned in 10.2 Days from an onset date of adverse events to the outcome confirmation date (recovered or recovering).

# "2.4.2 A list of the onset status of the priority survey items per 100 patient-year"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of the priority survey items per 100 patient-year by adverse event, serious adverse event, adverse reaction, serious adverse reaction of patients in the safety analysis group.

Analysis items: calculate the number of patients and the percentage to the number of patients in the analysis groups per type of seriousness and type of priority survey items for adverse events/reactions which occurred between the first administration date of Humira and the final administration date of Humira + 28.

In addition, calculate the number of events/reactions and the event rate per 100 patient-year.

Note: Aggregate the total number of developed events/reactions including the overlapped ones which occurred in a patient.

"2.5.1 A list of the onset status of adverse reactions with/without self-administration"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse reactions with/without self-administration Analysis item: aggregate the following items with/without self-administration for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, type of adverse reactions, etc. (SOC, PT).

"2.5.2 A list of the onset status of adverse reactions with/without self-administration"

Patients for analysis: patients excluded from the safety analysis group

Analysis objective: to show the onset status of adverse reactions with/without self-administration Analysis item: aggregate the following items with/without self-administration for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, type of adverse reactions, etc. (SOC, PT).

"2.6 Incidence of adverse reactions per onset period (serious)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of serious adverse reactions per the onset period.

Analysis item: aggregate the following items by period for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with serious adverse reactions, etc. number of serious adverse reactions, type of adverse reactions, etc. (SOC, PT).

Note: Aggregate the initial reactions among the identical PTs in a patient. Aggregate the events based on the segments which contain the initial onset period of adverse reactions among Time Allowance

defined in "12.4 Assessment period for the onset status of adverse reactions". When calculating the number of patients with the target reactions, remove overlapped data per case number and onset period. When calculating the number of SOC, remove the overlapped data per case number, onset period and SOC.

Count the number of target patients and reactions by using the dates defined below until the assessment period applicable to Time Allowance defined in "12.4 Assessment period for the onset status of adverse reactions".

- Discontinued patients: the final administration date of Humira + 28 days
- Not discontinued patients: the first administration date of Humira + 1120 days

Even if there is one adverse reaction, it should be counted as one patient in every period when the reaction persisted.

"2.7 Incidence of adverse reactions per set period"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse reactions per onset period.

Analysis item: aggregate the following items by period for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, type of adverse reactions, etc. (SOC, PT).

Note: Aggregate the initial reactions among the identical PTs in a patient. Aggregate the events based on the segments which contain the initial onset period of adverse reactions among Time Allowance defined in "12.4 Assessment period for the onset status of adverse reactions". When calculating the number of patients with the target reactions, remove overlapped data per case number and onset period. When calculating the number of SOC, remove the overlapped data per case number, onset period and SOC.

Count the number of target patients and reactions by using the dates defined below until the assessment period applicable to Time Allowance defined in "12.4 Assessment period for the onset status of adverse reactions".

- Discontinued patients: the final administration date of Humira + 28 days
- Not discontinued patients: the first administration date of Humira + 1120 days

Even if there is one adverse reaction, it should be counted as one patient in every period when the reaction persisted.

"2.9 Incidence of adverse reactions (serious adverse reactions/adverse reactions) per background factor"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the incidence of adverse reactions per patient background factor and analyze them.

Analysis items: calculate the number of all patients, the percentage to the number of patients with serious adverse reactions and all patients, the number of patients with adverse reactions and the percentage to number of all patients, the tests for adverse reactions (Fisher's exact test for nominal-scale factors and Man-Whitney's u test for ordinal-scale factors) per the following patient background factor regarding the adverse reactions which occurred in the safety analysis period. Note that the test does not include the patients "with treatment history with anti-TNF $\alpha$  drug for Crohn's disease".

Note: the patient background factors are as follows:

Sex, age (year), body weight (kg), BMI (kg/m<sup>2</sup>), duration of illness (year), indication (registration form), allergy history, smoking history, with smoking history (details), self-administration, tuberculosis test status, hepatitis B virus test status (registration form), complication; complication: liver disorder, complication: renal disorder, complication: blood disorder, complication: respiratory disorder, complication: diabetes mellitus, complication: osteoporosis, complication: malignant tumour, medical history, medical history: tuberculosis, medical history: non-tuberculous mycobacteriosis, medical history: interstitial pneumonia, medical history: bronchitis bacterial, medical history: aplastic anaemia, medical history: pancytopenia, medical history: malignant tumour, prior medication for Crohn's disease, prior medication: anti-TNFα drug, prior medication: aminosalicylic medication: acid drug, prior corticosteroids, prior medication: immunosuppressant, prior medication: antibiotics, prior treatment for Crohn's disease, prior treatment: surgery, prior treatment: GCAP, prior treatment: enteral nutrition therapy, prior treatment: intravenous nutrition therapy, treatment history with anti-TNFα drug for Crohn's disease, with treatment history with anti-TNFα drug for Crohn's disease, concomitant medication, concomitant medication: aminosalicylic acid drug, concomitant medication: corticosteroids, concomitant medication: immunosuppressant, concomitant medication: antibiotics, concomitant therapy for Crohn's disease, concomitant therapy: surgery, concomitant therapy: GCAP, concomitant therapy: enteral nutrition therapy, concomitant therapy; intravenous nutrition therapy, site of disease: anus/perianal region, site of disease: rectum, site of disease: stomach/duodenum, site of disease: colon, site of disease: jejunum/ileum, intestinal complication, non-intestinal complication, work condition, CDAI when the administration was started, CRP

"2.9.xx Incidence of adverse reactions per background factor and seriousness"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of non-serious/serious adverse reactions per statistically-significant background factor based on the test results in 2.9.

Analysis item: aggregate the following items per background factor and seriousness for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

"2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of non-serious/serious adverse reactions with/without hepatic function disorder

Analysis item: aggregate the following items with/without hepatic function disorder per seriousness regarding the adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

Note: Aggregate the most serious reaction among the identical PTs in a patient.

When calculating the number of patients with the target reactions, remove overlapped data per case number and seriousness. When calculating the number per SOC, remove the overlapped data per case number, seriousness and SOC.

"2.14.1 Incidence of adverse reactions with/without renal impairment and per seriousness"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of non-serious/serious adverse reactions with/without renal impairment

Analysis items: aggregate the following items with/without renal impairment per seriousness regarding the adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness".

"2.15.1 Incidence of adverse reactions per seriousness in pediatrics and non-pediatrics"

Patients for analysis: patients in the safety analysis group

Analysis objective: to separately show the onset status of serious or non-serious adverse reactions in pediatrics and non-pediatrics.

Analysis items: aggregate the following items per seriousness in pediatrics and non-pediatrics

regarding adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness".

"2.16.1 Incidence of adverse reactions per seriousness in the elderly and non-elderly patients" Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of non-serious/serious adverse reactions in the elderly and non-elderly patients.

Analysis items: aggregate the following items per seriousness in the elderly and non-elderly patients regarding adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness".

"2.17.1 A list of the onset status of adverse reactions/infections in this survey"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse reactions and serious adverse reactions.

Analysis item: aggregate adverse reactions and serious adverse reactions regarding the following items based on the adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, incidence of adverse reactions, etc., and type of adverse reactions, etc. (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness" for serious adverse reactions.

Put \* before the PT of unexpected events from "Precautions".

"2.17.2 A list of the onset status of adverse reactions/infections not in the follow-up period" Patients for analysis: patients whose survey form was locked

Analysis objective: to show the onset status of adverse reactions and serious adverse reactions which occurred not in the follow-up period.

Analysis item: aggregate adverse reactions and serious adverse reactions regarding the following

items based on the adverse reactions which occurred not in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, incidence of adverse reactions, etc., and type of adverse reactions, etc. (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness" for serious adverse reactions.

Put \* before the PT of unexpected events from "Precautions".

"2.17.3 A list of the onset status of adverse reactions/infections in this survey (patients excluded from the safety analysis)"

Patients for analysis: patients excluded from the safety analysis group

Analysis objective: to show the onset status of adverse reactions and serious adverse reactions.

Analysis item: aggregate adverse reactions and serious adverse reactions regarding the following items based on the adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, incidence of adverse reactions, etc., and type of adverse reactions, etc. (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness" for serious adverse reactions.

Put \* before the PT of unexpected events from "Precautions".

"2.19 A list of the onset status of adverse events in this survey"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse events, serious adverse events and non-serious adverse events.

Analysis items: aggregate adverse events, serious adverse events and non-serious adverse events regarding the following items among adverse events which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, number of adverse reactions, incidence of the reactions, type of adverse events (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness" for serious adverse events.

"2.20 A list of the onset status of adverse reactions (all cases)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the summary statistics on the days to the onset as well as the number of

patients per outcome and the days to the confirmed outcome (recovered or recovering) for adverse reactions.

Analysis items: calculate the number of cases and the percentage to the number of patients in the analysis groups per type of adverse reactions (SOC, PT), the number of patients with non-serious reactions and the percentage to the number of patients in the analysis groups, and the number of patients with serious reactions and the percentage to the number of patients in the analysis groups for the adverse reactions which occurred in the safety analysis period. In addition, calculate the summary statistics (the number of patients, the mean, the minimum, the median, the maximum) for days to the onset per PT, the number of patients per period from the onset date to the outcome (recovered or recovering), and the number of patients per outcome.

Note: When more than one identical PT is found in a patient, aggregate seriousness, days to the onset, outcome and days to the outcome (recovered or recovering) as 1 patient (case) in the following manner.

- Seriousness priority: serious > non-serious
- Days to the onset: identify the days as mentioned in "10.2 days from the first administration date of Humira to the adverse-event onset date".
- Outcome: identify it as specified in 10.2 Outcomes of adverse events
- Days to outcome (recovered or recovering): identify the days as mentioned in 10.2 Days from an onset date of adverse events to the outcome confirmation date (recovered or recovering).

# 13.3. Effectiveness

"3.1 CDAI remission rate at the final assessment (CDAI<150)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the remission rate of CDAI at the final assessment

Analysis items: calculate the number of target patients, the percentage to the number of patients who achieved a remission at the final assessment and to the number of target patients, and the percentage to the number of patients who failed to achieve a remission and to the number of target patients.

Note: Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for Time Allowance of the final assessment periods.

"3.2.1.1 Changes in Crohn's disease activity index (CDAI) since the administration was started (Observed Case)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show changes in CDAI and CDAI at each assessment period.

Analysis items: Calculate the number of target patients, the mean and standard deviation of CDAI,

the mean and standard deviation of changes in CDAI for each assessment period, and conduct a paired-t test which compares the values at the initial administration. In addition, calculate the mean days from the first administration date to the final assessment date and the  $\pm$  standard deviation.

Note: Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for Time Allowance of the final assessment periods. The analysis covers only the patients with the assessment at the first administration and thereafter.

"3.2.1.2 Changes in Crohn's disease activity index (CDAI) since the administration was started (Observed Case)"

Patients for analysis: the patients in the effectiveness analysis group whose CDAI was a remission (≥150) after they were started on Humira.

Analysis objective: to show changes in CDAI and the CDAI at each assessment period of patients whose CDAI failed to achieve a remission when the administration was started.

Analysis items: Calculate the number of target patients, the mean and standard deviation of CDAI, the mean and standard deviation of changes in CDAI for each assessment period, and conduct a paired-t test which compares the values at the initial administration. In addition, calculate the mean days from the first administration date to the final assessment date and the ± standard deviation.

Note: Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for Time Allowance of the final assessment periods. The analysis covers only the patients with the assessment at the first administration and thereafter.

"3.2.2.1 Changes in the remission rate at each point (CDAI<150) (Observed Case)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the remission rate of CDAI at each assessment period.

Analysis item: Calculate the number of target patients, the percentage to the number of patients who achieved a remission and the number of target patients, 95%CI of the remission rate, and conduct a McNemar test for the first administration per assessment period.

Note: Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for Time Allowance of the final assessment periods. The analysis covers only the patients with the assessment at the first administration and thereafter.

For the confidence interval, use the Clopper-Pearson's confidence interval.

"3.2.2.3 Changes in the remission rate at each point (CDAI<150) (Observed Case)"
Patients for analysis: the patients in the effectiveness analysis group whose CDAI was a remission (≥150) after they were started on Humira.

Analysis objective: to show the remission rate of CDAI at each assessment period of patients whose CDAI failed to achieve a remission when the administration was started.

Analysis item: Calculate the number of target patients, the percentage to the number of patients who achieved a remission and the number of target patients, 95%CI of the remission rate, and conduct a McNemar test for the first administration per assessment period.

Note: Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for Time Allowance of the final assessment periods. The analysis covers only the patients with the assessment at the first administration and thereafter.

For the confidence interval, use the Clopper-Pearson's confidence interval.

"3.2.4.2 Endoscopy results during administration (small intestine: active phase/remission phase)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show endoscopy results (small intestine) at each assessment period.

Analysis item: Calculate the number of patients who did not undergo endoscopy, the number of patients who underwent endoscopy, the percentage to the number of patients in the active phase and the number of patients who underwent endoscopy, the percentage to the number of patients in the remission phase and the number of patients who underwent endoscopy, and the mean days from the endoscopy prior to administration to the first administration date of Humira.

Note: Follow "12.2 Assessment period for endoscopy results" for Time Allowance of assessment period. The analysis covers only the patients with the endoscopy assessment (small intestine) at the first administration and thereafter in the effectiveness analysis group.

"3.2.5.2 Endoscopy results during administration (large intestine: active phase/remission phase)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the endoscopy results (large intestine) at each assessment period.

Analysis item: Calculate the number of patients who did not undergo endoscopy, the number of patients who underwent endoscopy, the percentage to the number of patients in the active phase and the number of patients who underwent endoscopy, the percentage to the number of patients in the remission phase and the number of patients who underwent endoscopy, and the mean days from the endoscopy prior to administration to the first administration date of Humira.

Note: Follow "12.2 Assessment period for endoscopy results" for Time Allowance of assessment period. The analysis covers only the patients with the endoscopy assessment (large intestine) at the first administration and thereafter in the effectiveness analysis group.

"3.2.5.3 Endoscopy results during administration (remission phase in both small and large intestines)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show endoscopy results in the remission phase (for small and large intestines) Calculate the number of patients who underwent endoscopy (for small and large intestines), the number of patients whose small and large intestines in the remission phase, and the percentage to the patients who underwent endoscopy (for small and large intestines).

Note: Follow "12.2 Assessment period for endoscopy results" for Time Allowance of assessment period. The analysis covers only the patients with the data showing that endoscopy for small and large intestines was done on the same day at the first administration and thereafter in the effectiveness analysis group.

"3.2.6.2 Changes in WPAI:CD since the administration was started (Observed Case)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show WPAI at each assessment period.

Analysis items: Calculate the number of target patients and the summary statistics of WPAI for each assessment period, and conduct a paired-t test which compares the values at the initial administration.

Note: Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for Time Allowance of the final assessment periods. The analysis covers only the patients with the WPAI assessment at the first administration and thereafter in the effectiveness analysis group.

"3.2.7.2 Changes in CRP level since the administration was started (Observed Case)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show CPR levels at each assessment period.

Analysis items: Calculate the number of target patients and the summary statistics of CRP for each assessment period, and conduct a paired-t test which compares the values at the initial administration.

Note: Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for Time Allowance of the final assessment periods. The analysis covers only the patients with the CRP assessment at the first administration and thereafter in the effectiveness analysis group.

"3.2.7.3 Remission rate at the final assessment in patients who achieved a remission of CDAI at Week 4 of administration"

Patients for analysis: Patients in the effectiveness analysis group (the patients who did not achieve a remission (≥150) when the administration was started but achieved the remission (<150) at Week 4 of administration in CDAI)

Patients for analysis: to show the remission rate of CDAI at the final assessment regarding the patients who did not achieve a remission ( $\geq$ 150) when the administration was started but achieved the remission (<150) at Week 4 of administration.

Analysis items: calculate the number of target patients, the percentage to the number of patients who achieved a remission at the final assessment and the target patients, and the 95% confidence interval of the remission rate.

Note: The target patients need to have their CDAI measured at 3 time points or more, that is, at the first administration, Week 4 of administration and any point after Week 4 of administration and also have a record that they did not achieve a remission ( $\geq$ 150) at the first administration but achieved the remission (<150) at Week 4 of administration.

Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for Time Allowance of the assessment periods.

For the confidence interval, use the Clopper-Pearson's confidence interval.

"3.2.8 Subsequent changes in the conditions of patients with non-intestinal conditions observed at the first administration (Observed Case)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the conditions at each assessment period regarding non-intestinal conditions observed at the first administration.

Analysis item: Calculate the number of target patients, the percentage to the number of patients with the conditions and the number of target patients, and conduct a McNemar test for the first administration per assessment period.

Note: The analysis covers only the patients with the assessment at the first administration and thereafter as well as the patients with symptoms for each "arthritis/arthralgia", "iritis/uveitis", and "erythema nodosum/gangrenous abscess/aphthous stomatitis" at the first administration.

To analyze "with any of non-intestinal conditions", the patients with any symptom at each assessment period regarding any of the items answered as 'with a symptom' at the first administration are regarded as the patients with conditions. When a patient had multiple symptoms at the first administration, they should be regarded as "with conditions" if any of the symptoms persisted. Do not include in analysis the items in which no symptoms were observed at the first administration. (Do not include in the analysis a symptom which first developed at an assessment

period after the first administration, either)

Follow "12.1 Assessment period for CDAI, WPAI, CRP and non-intestinal conditions" for Time Allowance of the assessment periods.

# "3.4.1 Aggregation for effectiveness per patient background factor (CDAI)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the CDAI remission rate at the final assessment per patient background factor and analyze them.

Analysis items: For CDAI at the final assessment, calculate the number of patients, the percentage to the number of patients who failed to achieve a CDAI remission and the number of patients per background factor, the number of patients who achieved a CDAI remission and the percentage to the number of patients per background factor, and the tests for CDAI remission (Fisher's exact test for nominal-scale factors and Man-Whitney's u test for ordinal-scale factors) per patient background factor below. Note that the test does not include the patients "with treatment history with anti-TNF $\alpha$  drug for Crohn's disease".

Note: the patient background factors are as follows:

Sex, age (year), body weight (kg), BMI (kg/m<sup>2</sup>), duration of illness (year), indication (registration form), allergy history, smoking history, with smoking history (details), self-administration, tuberculosis test status, hepatitis B virus test status (registration form), complication; complication: liver disorder, complication: renal disorder, complication: blood disorder, complication: respiratory disorder, complication: diabetes mellitus, complication: osteoporosis, complication: malignant tumour, medical history, medical history: tuberculosis, medical history: non-tuberculous mycobacteriosis, medical history: interstitial pneumonia, medical history: bronchitis bacterial, medical history: aplastic anaemia, medical history: pancytopenia, medical history: malignant tumour, prior medication for Crohn's disease, prior medication: anti-TNF $\alpha$  drug,prior medication: aminosalicylic acid drug, prior medication: corticosteroids, prior medication: immunosuppressant, prior medication: antibiotics, prior treatment for Crohn's disease, prior treatment: surgery, prior treatment: GCAP, prior treatment: enteral nutrition therapy, prior treatment: intravenous nutrition therapy, treatment history with anti-TNFα drug for Crohn's disease, with treatment history with anti-TNFα drug for Crohn's disease, concomitant medication, concomitant medication: aminosalicylic acid drug, concomitant medication: corticosteroids, concomitant medication: immunosuppressant, concomitant medication: antibiotics, concomitant therapy for Crohn's disease, concomitant therapy: surgery, concomitant therapy: GCAP, concomitant therapy: enteral nutrition therapy, concomitant therapy: intravenous nutrition therapy, site of disease: anus/perianal region, site of disease: rectum, site of disease: stomach/duodenum, site of disease: colon, site of disease: jejunum/ileum, intestinal complication, non-intestinal complication, work condition, CDAI when the administration was started, CRP